CLINICAL TRIAL: NCT07291323
Title: A Phase 1, Open-Label Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of JANX011 With Optional Step-Up Dosing in Healthy Adult Volunteers
Brief Title: Study of JANX011 in Healthy Adult Volunteers to Assess Safety and Tolerability.
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janux Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARMV-011-001
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Autoimmune

STUDY DESIGN:
Intervention Model Description: Subjects will receive one dose of JANX011 subcutaneously. Dosage per cohort will increase to determine the maximum tolerable dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Dosage per cohort will increase to determine the maximum tolerable dose.
  Interventions: Drug: JANX011

INTERVENTIONS:
Drug: JANX011 — JANX011 is administered subcutaneously, one time.

SUMMARY:
This first-in-human (FIH) study aims to characterize the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of JANX011 dosed subcutaneously (and potentially intravenously) in healthy adult volunteers (HVs) to gain insight into its therapeutic utility in patients with autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, in the opinion of the PI or designee and as determined by physical examination, laboratory screening tests, and medical history.
* Aged 18 to 65 years, with a body weight between 50 to 120 kg and a body mass index (BMI) between 18 to 32 kg/m2 (all inclusive) at Screening.
* Able and willing to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.

Exclusion Criteria:

* Recent surgery requiring general anesthesia within 12 weeks prior to Screening or is expected to have surgery requiring general anesthesia during the course of the study.
* Positive test for hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg), human immunodeficiency virus 1 (HIV-1) or HIV-2 antibodies.
* Positive test for tuberculosis (TB) or history of TB (including prior positive interferon gold test result).
* Use of any investigational medical device or investigational drug within 30 days or 5 half-lives of the investigational drug (whichever is longer) prior to dosing on Day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, and relatedness of TEAEs, treatment-emergent SAEs, and treatment-emergent AESIs. | Up to 85 days

CONTACTS AND LOCATIONS:
Overall Officials: Zach McIver, D.O., PhD, Study Chair — Janux Therapeutics
Locations (1):
- CMAX, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No